CLINICAL TRIAL: NCT03576521
Title: Efficacy of Ocoxin-Viusid in the Prevention of Acute Toxicity by Chemotherapy in Patients With Breast Cancer. Phase II Clinical Trial
Brief Title: Evaluation of Ocoxin®-Viusid® in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OOS-CANCER-11
Record Dates: First submitted 2018-06-13; First posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer; Breast Carcinoma; Adriamycin Toxicity; Cyclosporine Toxicity
Keywords: breast cancer; chemotherapy toxicity; Oxidative Stress; Nutritional supplement; Ocoxin Viusid
MeSH Terms: conditions — Breast Neoplasms | interventions — Ocoxin

STUDY DESIGN:
Intervention Model Description: Phase II randomized, controlled, double blind clinical trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: A double blind. The masking will be maintained until the analysis of the data. However, access to the code will be allowed if serious adverse events arise related to the research product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ocoxin-Viusid® (Experimental): The CT with Adriamycin 60 mg per m2 of Body Surface (BS) and Cyclophosphamide Infusion intravenous every 21 days, up to a total of 4 to 6 cycles + OV nutritional supplement.
  Interventions: Combination Product: CT + Ocoxin-Viusid
- Placebo (Placebo Comparator): The QT Adriamycin scheme 60 mg per m2 of Body Surface (SC) and Cyclophosphamide Infusion intravenous every 21 days, up to a total of 4 to 6 cycles + a placebo of the OV nutritional supplement.
  Interventions: Combination Product: CT + Placebo

INTERVENTIONS:
Combination Product: CT + Ocoxin-Viusid — The included patients received the Ocoxin-Viusid nutritional supplement at a rate of 75 ml daily (25 ml in 3 doses every 8 hours) administered after main meals diluted in milk or juice. The treatment will start a week before, it will be maintained throughout the coventional chemotherapy treatment* and up to three weeks after the end of the treatment.
  *All patients should receive the CT Adriamycin 60 mg per m2 of Body Surface (BS) and Cyclophosphamide Infusion intravenous every 21 days, up to a total of 4 to 6 cycles according to protocols provided in the center.
  Arms: Ocoxin-Viusid®
Combination Product: CT + Placebo — The included patients received the OV placebo in oral solution at a rate of 75 ml daily (25 ml in 3 doses every 8 hours), administered after main meals diluted in milk or juice. The treatment will start a week before, it will be maintained throughout the coventional chemotherapy treatment* and up to three weeks after the end of the treatment.
  *All patients should receive the CT Adriamycin 60 mg per m2 of Body Surface (BS) and Cyclophosphamide Infusion intravenous every 21 days, up to a total of 4 to 6 cycles according to protocols provided in the center.
  Arms: Placebo

SUMMARY:
The purpose is to determine the efficacy of the nutritional supplement Ocoxin-Viusid oral solution (OV) in the reduction of acute toxicity of Chemotherapy (CT) treatment with patients with breast carcinoma. A randomized, double-blind phase II clinical trial was designed, with a sample of 120 patients distributed in 2 arms: 60 patients will receive the CT treatment plus the OV, 60 will receive CT plus OV placebo. The OV / placebo will be administered before, during and 3 weeks after the conclusion of the CT. A better tolerance to the treatment is expected with the addition of the nutritional supplement.

DETAILED DESCRIPTION:
To obtain the sample size, the proportion of patients presenting adverse reactions that require interrupting chemotherapy treatment will be taken into account. In the institution, this figure is close to 15%. Since it is a dietary supplement, with extensive information on the safety of the product, the design is used in a stage of Flemming (without early stop rules). Assuming that the Ocoxin-Viusid product would clearly be declared ineffective (maximal ineffectiveness) if the proportion of patients not presenting adverse reactions was equal to less than 85% (p0), that is the maximum level of success below which the product does not shows signs of efficacy (the study does not guarantee further research) and taking a p1 value of 95%, where p1 is the minimum level of efficacy required from which the product would be declared effective (the results guarantee to continue a study phase III). Assuming an α error of 5% (probability of rejecting the null hypothesis when it is true) and β (probability of rejecting the alternative hypothesis when it is true) of 20% (the power of the test: 1 - β = 80%), It is determined to recruit a maximum number of 59 - 60 subjects. Determine a = 54, where a is the number of responses equal and below which the product is declared ineffective (H0 is accepted). And r = a + 1 is the cut-off point, that is, the number of responses from which the efficacy level ensures to continue to a phase III study. In this case we would expect to obtain a number of successes ≥ 55.

Patients will be randomized after surgery, in the chemotherapy consultation, and once they meet the established inclusion criteria. In order to achieve the masking of the research product, these have been labeled by a balanced randomized list obtained by computer, which will be in the possession of the Biostatistician of the study of the Clinical Investigations Section of INOR and the promoter. The product under study has been consecutively labeled from 1 to 120 (60 patients in each therapeutic arm).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone surgery and histologically confirm a breast carcinoma and who are subject to adjuvant treatment with AC chemotherapy at the time of inclusion in the trial.
2. Patients with age ≥18 years of female sex.
3. General health status according to the Karnofsky Index ≥ 70.
4. Laboratory parameters within the normal limits defined to receive this chemotherapy including normal Echocardiogram:

   to. Hematopoietic: Hemoglobin ≥ 9 g / L, Total Leukocytes ≥ 3 x 109 cells / L, Neutrophils ≥ 1.5 x 109 cells / L, Platelets ≥ 100 x 109 / L.

   b. Hepatic: Liver function within 2.5 times upper normal limit and without liver disease demonstrated by TGP, OGT and alkaline phosphatase.

   c. Renal function: creatinine ≤ 132 μmol / l.
5. Patients who express written voluntariness to enter the study with their signature of the informed consent document.
6. Patients of childbearing age with negative pregnancy test or who have effective contraceptive methods such as intrauterine devices, hormonal contraceptives, barrier method or tubal ligation.

Exclusion Criteria:

1. Patients who have received prior chemotherapy.
2. Patients who are receiving another research product.
3. Patients with known hypersensitivity to any ingredient of the investigational product.
4. Decompensated intercurrent diseases, including: active infections, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, hepatic diseases and psychiatric illnesses that could limit adherence to the requirements of the clinical trial or any other special condition that at the discretion of the physician put your health or life at risk during your participation in the trial.
5. Pregnancy, lactation or puerperium.
6. Patients with cerebral metastases and / or leptomeningeal carcinosis.
7. Patients with a second concomitant tumor.
8. Patients carrying the human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05-13 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
The Ocoxin-Viusid effect in the treatment with chemotherapy | 4 months
  The effect of the treatment will be evaluated from the number of interruptions of oncospecific treatment due to acute toxic reactions to chemotherapy.
Compliance with the planned chemotherapy schedule | 4 months
  Dichotomous variable that will be evaluated through the answer yes or no. In cases of negative response, the cause of non-compliance will be collected. It will be collected in the evaluation corresponding to each cycle of chemotherapy and in the final evaluation.
The Ocoxin-Viusid effect in the treatment with chemotherapy | 4 months
  The effect of the treatment will be evaluated from the percentage of interruptions of oncospecific treatment due to acute toxic reactions to chemotherapy.

SECONDARY OUTCOMES:
Evaluation of Quality of Life | 4 months
  It will be measured through the Karnofsky Index. The Karnofsky Index will be collected in each evaluation query (score of 0-100 points at intervals of 10).
Evaluation of Quality of Life | 4 months
  It will be measured through quality of life scale of the EORTC QLQ-C30 (general). It's a questionnaire of 30 questions divided into 3 areas: Functional capacity (physical aspect, social role, cognitive capacity, emotional and social factors; yes or no), symptoms (asthenia, pain and nausea / vomiting; from 1 to 4) and global assessment (from 1 to 10)
Evaluation of Quality of Life | 4 months
  It will be measured through quality of life scale of the EORTC QLQ-BR23 (specific for breast cancer), it contains 31-53 questions, with a scale from 1-4 or 1-7 (bad-excellent):
  -Functional scales:
  Body image (BRBI) Sexual functioning (BRSEF) Sexual enjoyment (BRSEE) Future perspective (BRFU)
  -Symptom scales / items
  Systemic therapy side effects (BRST) Breast symptoms (BRBS) Arm symptoms (BRAS) Upset by hair loss (BRHL)
Evaluation of nutritional status | 4 months
  It will be determined through the Body Mass Index (BMI). The investigator must take into account that if the patient presents with ascites, she should indicate a paracentesis (whenever possible and the type of ascites allows it) before measuring her body weight.
Evaluation of nutritional status | 4 months
  It will be determined through the value of total proteins and albumin.
Side effects of the treatment | 4 months
  The safety of the treatment will be determined through the reporting of adverse events that are presented to the research product.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Oncology and Radiobiology (INOR), La Habana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR